CLINICAL TRIAL: NCT00037479
Title: PET and MRI Imaging of Persistent Lyme Encephalopathy
Brief Title: Brain Imaging and Retreatment Study of Persistent Lyme Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: R01NS038636 (NIH)
Record Dates: First submitted 2002-05-17; First posted 2002-05-20 (Estimated); Last update posted 2005-12-07 (Estimated); Status verified 2005-12

CONDITIONS: Lyme Disease; Lyme Neuroborreliosis
Keywords: neurologic Lyme disease; Lyme disease; ceftriaxone; Rocephin; PET scans; Lyme encephalopathy; neuroborreliosis; borreliosis
MeSH Terms: conditions — Lyme Disease; Lyme Neuroborreliosis; Borrelia Infections | interventions — Ceftriaxone

INTERVENTIONS:
Drug: ceftriaxone

SUMMARY:
The purpose of this study is to determine whether patients with persistent memory problems after Lyme disease benefit from an additional longer course of IV antibiotic therapy; to use modern brain imaging technology to determine whether the problem in the central nervous system is primarily one of poor blood flow or one of impaired nerve cell functioning; and to try to identify biological markers prior to treatment that will identify patients who are more or less likely to respond to the study treatment.

DETAILED DESCRIPTION:
Some people with a history of Lyme disease continue to have problems despite having received "textbook duration" antibiotic therapy. When memory, attention, or thinking problems persist, the syndrome is called persistent Lyme disease (PLD). This study seeks to answer critical scientific questions about the treatment and cause of PLD symptoms.

This 24-week treatment study will evaluate each patient's response to treatment using neuropsychological testing and state-of-the-art brain imaging. The brain tests include neuropsychological testing of memory and attention, brain imaging (MRI and PET scans) to look at blood flow in the brain and nerve cell structure and metabolism, a neurological exam, and studies of the fluid that surrounds the brain (cerebrospinal fluid). The treatment involves 10 weeks of either intravenous antibiotic called ceftriaxone (also known as Rocephin) or intravenous placebo (inactive substance). After the first visit to Columbia Presbyterian Medical Center, the remaining treatments will be done in the patient's home. Patients will be screened over the phone and in person to confirm study eligibility.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants must:

* Be 18-65 years old
* Have persistent problems with memory, verbal fluency, or attention after having contracted Lyme disease.
* Be able to travel to New York for 4-5 evaluations over the course of one year. Travel costs for participants in need may be partially or fully reimbursable.
* Have had a history of well-documented Lyme disease using the CDC's clinical criteria and a current positive IgG Western blot or PCR.
* Have received, at some point in the past at least 3 weeks of IV antibiotic therapy for Lyme disease.

Exclusion Criteria:

Ineligible from participation are people with the following:

* Other major medical or neurologic problems
* Smoke more than 10 cigarettes a day
* Uncontrolled high blood pressure
* Allergy to ceftriaxone (Rocephin)
* History of marked cocaine abuse

Twenty healthy subjects are also being sought for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65
Dates: Start 1999-12

CONTACTS AND LOCATIONS:
Overall Officials: Brian Fallon, M.D., Principal Investigator — Columbia University, College of Physicians and Surgeons, Lyme Disease Research Program
Locations (1):
- Columbia Presbyterian Medical Center, New York, New York, United States

REFERENCES:
- See also: Columbia's Lyme disease research studies website — http://www.columbia-lyme.org